CLINICAL TRIAL: NCT03249116
Title: Assessing Mechanisms of Anxiety Reduction in Animal-assisted Interventions for Adolescents With Social aAnxiety
Brief Title: Assessing Mechanisms of Anxiety Reduction in Animal-assisted Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Megan K Mueller, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R03HD091892-01 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Social Anxiety Disorder; Social Anxiety; Social Anxiety Disorder of Childhood
Keywords: human-animal interaction; animal-assisted intervention
MeSH Terms: conditions — Phobia, Social; Human-Animal Interaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control - interaction with a stuffed dog (Active Comparator): Active control - interaction with a stuffed dog
  Interventions: Other: active control
- Therapy dog - social (Experimental): animal-assisted intervention - social interaction only with therapy dog during stress task.
  Interventions: Other: animal-assisted intervention
- Therapy dog - Social + physical (Experimental): animal-assisted intervention - Social interaction and physical interaction with therapy dog during stress task.
  Interventions: Other: animal-assisted intervention

INTERVENTIONS:
Other: animal-assisted intervention — Interaction with a therapy dog
  Arms: Therapy dog - Social + physical; Therapy dog - social
Other: active control — Interaction with a stuffed dog
  Arms: Control - interaction with a stuffed dog

SUMMARY:
Adolescence and young adulthood is a critical period for the development of social anxiety, which is often linked to other mental health challenges such as depression, mood disorders, and substance abuse. Initial evidence suggests that interacting with animals can reduce stress and anxiety, but no research has tested whether this benefit extends to adolescents at risk for social anxiety disorder. Additionally, researchers and clinicians do not understand what mechanism is responsible for anxiety reduction in animal-assisted interventions (AAIs). Therefore, the objectives of this study are to explore the specific mechanisms by which interacting with a therapy dog reduces anxiety, and to test whether such an interaction reduces anxiety in adolescents with varying levels of social anxiety.

DETAILED DESCRIPTION:
The specific aims of this project are to (1) test the mechanisms by which AAIs reduce anxiety, and (2) determine if the anxiolytic effect of social and physical interaction is moderated by level of pre-existing social anxiety. To achieve these aims, 75 adolescents (age 13-17) will undergo a well-validated laboratory-based social evaluative stressor, the Trier Social Stress Task for Children, and be randomly assigned to one of three conditions: 1) no interaction with a dog (control condition), 2) social interaction only (no physical interaction) with a therapy dog; or 3) social interaction plus physical interaction with a therapy dog. Using a multivariate approach, three levels of outcome data will be collected: a) self-reported experience (anxiety), b) autonomic physiology (heart rate), and c) behavioral performance (error rates on mental math task). In addition, the interactions will be videotaped and behavioral coding will be used to explore the specific social behaviors between the participant and the dog that may predict anxiety reduction (such as frequency or type of social referencing or physical contact).

ELIGIBILITY:
Inclusion Criteria:

- Low, mid-range, and high levels of social anxiety

Exclusion Criteria:

* Fear of dogs
* Allergy to dogs

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan K Mueller, PhD, Principal Investigator — Tufts University
Locations (1):
- Cummings School of Veterinary Medicine at Tufts University, North Grafton, Massachusetts, United States

REFERENCES:
- [Derived] Mueller MK, Anderson EC, King EK, Urry HL. Null effects of therapy dog interaction on adolescent anxiety during a laboratory-based social evaluative stressor. Anxiety Stress Coping. 2021 Jul;34(4):365-380. doi: 10.1080/10615806.2021.1892084. Epub 2021 Mar 2. PMID 33650444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 75 adolescents ages 13-17 on a continuum of social anxiety who were recruited through convenience and snowball sampling via local libraries and youth centers, social media, and other public venues.
Groups:
- Control: Active control - interaction with a stuffed dog only
- Therapy Dog - Social: animal-assisted intervention - social interaction only with therapy dog during TSST.
  animal-assisted intervention: Interaction with a therapy dog
- Therapy Dog - Social + Physical: animal-assisted intervention - Social interaction and physical interaction with therapy dog during TSST.
  animal-assisted intervention: Interaction with a therapy dog
Period: Overall Study
Arm/Group | Control | Therapy Dog - Social | Therapy Dog - Social + Physical
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Interaction With a Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 25 | 75
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.4) | 15.4 (1.6) | 15.7 (1.4) | 15.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 7 | 46
  Male | 8 | 3 | 18 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 25 | 23 | 23 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 22 | 23 | 20 | 65
  More than one race | 0 | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 25 | 75
Social anxiety level [Count of Participants; unit: Participants]
  Low Anxiety | 8 | 6 | 4 | 18
  Mid Anxiety | 7 | 6 | 9 | 22
  High Anxiety | 10 | 13 | 12 | 35
Pet ownership [Count of Participants; unit: Participants] | 19 | 17 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Affective Experience
Description: The state scale of the State-Trait Anxiety Inventory (STAI) was used to measure state-level anxiety. We used the six-item short form of the STAI, which asks participants to rate how each of the six words reflects their feelings (calm, upset, relaxed, worried, tense, content). The short form was originally administered as a four-point scale, which we further modified to a three-point scale for feasibility in administering repeatedly over a short time period (response options for each item followed the format: very calm, calm, not calm). Responses to the six items were used to create a sum score at each time point with a possible range of 3 to 18 (higher scores indicate higher levels of anxiety).
Time Frame: Self-reported anxiety was measured at six time points, during: (Time 1; 0 min) baseline, (Time 2; 30 min) anticipation, (Time 3; 35 min) preparation, (Time 4; 45 min) speech, (Time 5; 60 min) recovery period 1, and (Time 6; 75 min) recovery period 2.
Population: 7 participants were excluded due to protocol deviations (not following study directions), and 2 had missing data for self-reported affective experience.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control - Stuffed Dog: active control: Interaction with a stuffed dog
Arm/Group | Control - Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical
Number analyzed (Participants) | 21 | 20 | 25
units on a scale
  Time 1 - 0 min | 10.19 (1.81) | 10.00 (2.07) | 10.28 (1.60)
  Time 2 - 30 min | 8.33 (1.88) | 8.05 (1.32) | 7.88 (1.67)
  Time 3 - 35 min | 12.05 (2.01) | 11.96 (2.44) | 12.36 (2.18)
  Time 4 - 45 min | 13.57 (2.40) | 13.14 (2.32) | 13.40 (2.40)
  Time 5 - 60 min | 9.33 (1.53) | 9.14 (1.93) | 8.68 (2.51)
  Time 6 - 75 min | 8.43 (1.43) | 8.52 (1.44) | 8.72 (2.01)
Statistical Analysis 1: Comparison: Control - Stuffed Dog vs Therapy Dog - Social vs Therapy Dog - Social + Physical; Test type: Superiority; p = .723, ANOVA — The threshold for statistical significance was p<.05; dependent variable: self-reported anxiety between-subjects factors: condition, social anxiety within-subjects factor: time; F statistic = 0.33

2. Secondary Outcome: Autonomic Physiological Reactivity: Electrodermal Activity
Description: Electrodermal activity (EDA) was recorded at 4 Hz by an Empatica E4 wristband sensor. EDA is reported in μSiemens with higher values representing higher levels of autonomic reactivity. EDA was recorded continuously, and for analysis was assessed over six time windows during the experiment: Time 1 = beginning of study; Time 2 = baseline period; Time 3 = anticipation phase; Time 4 = last 5 min of the stressor; Time 5 = recovery 1; Time 6 = recovery 2. Each time point was 5 minutes in duration.
Time Frame: Continuous through the 2 hour experiment.
Population: 7 participants were excluded for having a protocol deviation and 14 participants with EDA data that were not usable (3 of whom also had a protocol deviation)
Measure: Mean (Standard Deviation); unit: μSiemens
Groups:
- Control - Stuffed Dog: Active control - interaction with a stuffed dog
Arm/Group | Control - Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical
Number analyzed (Participants) | 17 | 20 | 20
μSiemens | 7.32 (3.03) | 6.56 (2.52) | 8.01 (3.41)
Statistical Analysis 1: Comparison: Control - Stuffed Dog vs Therapy Dog - Social vs Therapy Dog - Social + Physical; Test type: Superiority; p = .271, ANOVA — The threshold for statistical significance was p<.05; dependent variable: electrodermal activity between-subjects factors: condition, social anxiety within-subjects factor: time; F statistic = 1.34

3. Secondary Outcome: Autonomic Reactivity: Heart Rate
Description: Heart rate (beats per minute) Heart rate was measured via photoplethysmography from the Empatica E4 wristband using Empatica's proprietary algorithm, which automatically imputes missing data from the photoplethysmograph signal and corrects for motion artifacts. The heart rate is computed as the average heart rate values that spans 10 seconds. This average HR is computed at 1 Hz. HRwas recorded continuously, and for analysis was assessed over six time windows during the experiment: Time 1 = beginning of study; Time 2 = baseline period; Time 3 = anticipation phase; Time 4 = last 5 min of the stressor; Time 5 = recovery 1; Time 6 = recovery 2. Each time point was 5 minutes in duration.
Time Frame: continuous through the 2 hour experiment
Population: 7 participants were excluded due to protocol deviations (not following study directions).
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Control - Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical
Number analyzed (Participants) | 21 | 22 | 25
Beats per minute | 79.48 (7.92) | 78.73 (10.55) | 80.44 (11.36)
Statistical Analysis 1: Comparison: Control - Stuffed Dog vs Therapy Dog - Social vs Therapy Dog - Social + Physical; Test type: Superiority; p = .638, ANOVA — The threshold for statistical significance was p<.05; dependent variable: heart rate between-subjects factors: condition, social anxiety within-subjects factor: time; F statistic = 0.45

4. Secondary Outcome: Cognitive Performance - Number of Errors
Description: Number of errors (incorrect answer to subtraction task) during mental math task; better performance was characterized by fewer errors. Number of errors ranged from 0 to 8.
Time Frame: 1 hour into 2 hour experiment
Population: 7 participants were excluded due to protocol deviations (not following study directions).
Measure: Mean (Standard Deviation); unit: number of errors
Arm/Group | Control - Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical
Number analyzed (Participants) | 21 | 22 | 25
number of errors | 3.29 (1.95) | 3.36 (2.24) | 3.20 (2.20)
Statistical Analysis 1: Comparison: Control - Stuffed Dog vs Therapy Dog - Social vs Therapy Dog - Social + Physical; Test type: Superiority; p = .868, ANOVA — The threshold for statistical significance was p<.05; dependent variable: number of errors between-subjects factors: condition, social anxiety; F statistic = 0.14

5. Secondary Outcome: Cognitive Performance - Lowest Number Reached/Highest Number of Correct Responses
Description: Highest number of correct responses in serial subtraction task. To adjust for the different levels of subtraction based on age level, lowest number reached was operationalized by calculating the number of correct responses (a higher score indicating better performance). Number of correct answers ranged from 1 to 41.
Time Frame: 1 hour into 2 hour experiment
Population: 7 participants were excluded due to protocol deviations (not following study directions)
Measure: Mean (Standard Deviation); unit: highest number of correct responses
Arm/Group | Control - Stuffed Dog | Therapy Dog - Social | Therapy Dog - Social + Physical
Number analyzed (Participants) | 21 | 22 | 25
highest number of correct responses | 12.95 (8.85) | 13.41 (9.48) | 14.92 (12.59)
Statistical Analysis 1: Comparison: Control - Stuffed Dog vs Therapy Dog - Social vs Therapy Dog - Social + Physical; Test type: Superiority; p = .809, ANOVA — The threshold for statistical significance was p<.05; dependent variable: lowest number reached/highest number of correct responses between-subjects factors: condition, social anxiety; F statistic = 0.21

ADVERSE EVENTS:
Time Frame: 75 minutes
Description: Adverse events systematically collected for each participant via a standardized recording sheet. No adverse events occurred.
Groups:
- Control: Active control - interaction with a therapy dog
  active control: Interaction with a stuffed dog
Arm/Group | Control | Therapy Dog - Social | Therapy Dog - Social + Physical
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Heart rate data was of poor quality due to movement artifacts and therefore unable to be reliably interpreted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03249116/Prot_000.pdf
  • Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03249116/ICF_001.pdf
  • Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03249116/SAP_002.pdf